CLINICAL TRIAL: NCT04888754
Title: A Prospective Cohort for ex Vivo Cure Studies With Chronic HIV Infected Patients in the Netherlands: The CHRONO Project
Brief Title: A Prospective Cohort for ex Vivo Cure Studies With Chronic HIV Infected Patients in the Netherlands
Acronym: CHRONO
Status: Active, not recruiting | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Casper Rokx, Principal Investigator, Erasmus Medical Center
Other Study IDs: NL72765.078.20
Record Dates: First submitted 2021-04-14; First posted 2021-05-17 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: HIV Infections; HIV-1-infection; HIV-2 Infection
Keywords: HIV; HIV cure; HIV reservoir
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples and leucapheresis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A prospective non-interventional cohort study at Erasmus MC of adult chronic HIV infected patients of ≥18 years of age who initiate antiretroviral therapy in routine care.

DETAILED DESCRIPTION:
HIV cannot be cured with the current treatment armamentarium. A reservoir of latently HIV infected long lived CD4+T-cells is present in patients with HIV that are not affected by antiretroviral therapy. The evolution of this reservoir after therapy initiation is ill understood, as are the potential strategies to eradicate this reservoir. This study aims to anticipate on future HIV cure strategies by building a cohort to study ex vivo the reservoirs of HIV patients, the obstacles to cure HIV, and new therapeutic compounds and strategies.

Main study parameters/endpoints:

1. Change in viral reservoir size after antiretroviral treatment initiation.
2. Evolution of phenotypical and functional aspects of the anti-HIV host immune responses.
3. Ex vivo activity of established and novel HIV latency reversing agents.
4. Variance in HIV reservoir and host immunity between HIV subtypes and clinical variables.

A project from the Erasmus MC HIV Eradication Group (EHEG).

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years.
* Confirmed HIV-1 or HIV-2 infection
* Judged willing to initiate and adhere to cART by the HIV physician.

Exclusion Criteria:

* Inability to place venous catheters to draw blood.
* Major comorbidities:

  1. Severe symptomatic anemia or recent symptomatic cardiovascular event (un-stable angina pectoris, decompensated heart failure, myocardial infarction).
  2. The inability to participate due to any other relevant social, environmental,psychological, factors or according to the HIV treating physician's judgement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are 18 years or older with a confirmed HIV infection without prior exposure to cART (treatment naïve). Prior use of pre-exposure prophylaxis is allowed.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2021-05-26 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2034-01 (Estimated)

PRIMARY OUTCOMES:
To develop a prospective cohort in the Netherlands of chronic HIV infected patients within-depth reservoir characterization for future cure interventions. | 5-10 years
  The HIV latent reservoir will be characterised in chronic HIV patients using novel techniques like FISH-flow
To study the evolution of the HIV reservoir and immune host responses over time during antiretroviral therapy. | 5-10 years
  The HIV reservoir will be characterised over time to study the dynamics of the reservoir

SECONDARY OUTCOMES:
To explore established and putative new interventions aimed at curing HIV. | 5-10 years
  Blood and leucapheresis samples will be collected for testing of HIV cure drugs
To explore differences in reservoir size, activity and host responses, and their relation with clinical characteristics, between patients with different dominant HIV subtypes and sexes. | 5-10 years
  Blood and leucapheresis samples will be collected for reservoir characterisation to compare reservoirs between patients
To compare and validate new reservoir assays with current established assays. | 5-10 years
  Blood and leucapheresis samples will be collected to compare and validate new reservoir assays

CONTACTS AND LOCATIONS:
Overall Officials: Casper Rokx, MD PhD, Principal Investigator — Erasmus Medical Center; Tokameh Mahmoudi, PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus MC, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
No definitive decision on this yet. This will also depend on confidentiality.